CLINICAL TRIAL: NCT05969652
Title: Comparison of the Effectiveness of Supervised Heavy Slow Resistance Training and Eccentric Exercise Training in Patients With Rotator Cuff Tendinopathy: A Randomized Controlled Clinical Trial
Brief Title: Comparison of the Effectiveness Heavy Slow Resistance and Eccentric Training in Rotator Cuff Tendinopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Dilek Hande Esen, MSc, PT, Principal Investigator, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-77082166-302.08.01-547254
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Rotator Cuff Tendinopathy; Subacromial Impingement Syndrome; Bicep Tendinitis
Keywords: Exercise therapy; Rehabilitation; Resistance training; Shoulder pain; Subacromial impingement syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Two groups will be treated. The first group (experimental group) will be called the heavy slow resistance (HSR) group. The second group (control group) will be called the eccentric exercise (EE) group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not know which group they belong to. Doctors examining patients will also be blinded to group information. Which group the patients are included in will be the primary investigator who only performs the exercises.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heavy slow resistance group (HSR group) (Experimental): The investigators are planning a 6-week rehabilitation program, 2 days a week. The same physiotherapy and home exercise program will be applied to both groups. The physiotherapy and home exercise program will include patient education, stretching, range of motion and posture exercises. Resistance training will consist of different exercise principles but the same types of exercises. Resistance training: Dumball will be used as exercise equipment. Exercise intensity determined using the Numerical Pain Rating Scale (NPRS).
  Individual loading will be made according to the amount of weight. The maximum amount of pain producing pain less than 4 on the Numerical Pain Assessment Scale will be determined as exercise intensity. It will include 3 different exercises: 1) Full can. 2) External rotation in side lying. 3) Internal rotation in side lying.
  Interventions: Other: Heavy slow resistance training
- Eccentric exercise training group (EE group) (Active Comparator): The investigators are planning a 6-week rehabilitation program, 2 days a week. The same physiotherapy and home exercise program will be applied to both groups. The physiotherapy and home exercise program will include patient education, stretching, range of motion and posture exercises. Resistance training will consist of different exercise principles but the same types of exercises. Resistance training: Dumball will be used as exercise equipment. Exercise intensity determined using the Numerical Pain Rating Scale (NPRS).
  Individual loading will be made according to the amount of weight. The maximum amount of pain producing pain less than 4 on the Numerical Pain Assessment Scale will be determined as exercise intensity. It will include 3 different exercises: 1) Full can. 2) External rotation in side lying. 3) Internal rotation in side lying.
  Interventions: Other: Eccentric exercise training

INTERVENTIONS:
Other: Heavy slow resistance training — Patients will perform the exercises in the concentric and eccentric phases with the maximum amount of weight tolerated at a rate of 3 seconds/repetition. The number of sets*repetitions is given below. 2-3 minutes rest between sets will be given.
  1st week 3*15 2-3.week 3*12 4th-5th week 3*10 6th week 3*8
  Arms: Heavy slow resistance group (HSR group)
Other: Eccentric exercise training — Among the patients in the eccentric exercise group, only the eccentric phase of the exercises in the HSR group, will be asked to actively engage with the affected party. The eccentric contraction rate will be set to 6 seconds. Each exercise will be done 3 sets of 15 repetitions. In the next week, progress will be made in exercise intensity according to tolerance and 500 g will be added to the previous weight.
  will be continued. If patients cannot tolerate the new weight or there is an increase in pain, the same weight will be continued for another week.
  Arms: Eccentric exercise training group (EE group)

SUMMARY:
Rotator cuff tendinopathy, also called subbracromial impingement syndrome, is one of the most important causes of anterior shoulder pain. Although exercise training is known as an effective intervention method in the treatment of rotator cuff/subacromial impingement problems, there is no definite consensus on which type of exercise is more effective. The aim of this study is to analyze and compare the effects of the Heavy Slow Resistance (HSR) training and eccentric exercise training on pain, function, supraspinatus tendon structure, muscle strength, range of motion, subjective perception of improvement and treatment satisfaction in individuals with subacromial shoulder pain associated with rotator cuff tendinopathy.

DETAILED DESCRIPTION:
Rotator cuff tendinopathy, also called subbracromial impingement syndrome, is one of the most important causes of anterior shoulder pain. The most frequently affected structure in rotator cuff tendinopathies is the supraspinatus tendon due to its position in the subacromial space. Histological examinations of rotator cuff tendinopathy revealed that the structural changes in supraspinatus tendon injuries are similar to those of the patella and Achilles tendon injuries.

In the treatment of Achilles and patellar tendinopathy, it has been shown that eccentric exercise training has positive effects on pain and function, and supports the improvement in the structural and mechanical properties of the tendon. This success of eccentric training in managing lower extremity tendinopathies has encouraged researchers to conduct more scientific studies to develop evidence-based eccentric training guidelines for the conservative treatment of tendinopathies in the shoulder region. Studies showing that eccentric exercise training has positive effects on pain and function in rotator cuff pathologies have begun to take their place in the literature. In some studies, it has been stated that eccentric exercises are a safe and tolerable approach even in patients with rotator cuff tendinopathy who are candidates for arthroscopic subacromial decompression surgery and reduce the number of patients who are candidates for surgery. Again, in a systematic review-meta-analysis study involving individuals with rotator cuff tendinopathy, it was once again summarized that eccentric training has positive effects on pain and function, but it was stated that more studies are needed on this subject.

The HSR training is the repetitive gradual and slow contraction of the muscle against the heaviest possible load that the person can tolerate. In this training, the focus is more on the concentric and eccentric phases of the movement, and these phases are requested to be completed slowly in 3 seconds. As a result, the concentric/eccentric phase of an exercise repetition is performed with maximum weight in 6 seconds in total. There is scientific evidence in the current literature that slow resistance training has positive effects on symptoms and tendon structure in patella and Achilles tendinopathy. Beyer et al. compared eccentric exercise training and HSR training in Achilles tendinopathy and reported that both trainings had equally positive effects. However, scientific studies investigating the effects of slow resistance training in rotator cuff pathologies are mostly new and few in number. In a recent single-blind randomized controlled feasibility study conducted on 22 individuals with rotator cuff-related subacromial shoulder pain, the effects of slow resistance training in addition to traditional physical therapy program and traditional physical therapy program were compared. Schydlowsky et al. In their study comparing the effects of a supervised and home-based physiotherapy program in subacromial impingement syndrome, they did not directly examine the effects of slow resistance training, but used the slow resistance training procedure for the rotator cuff muscles.

Although exercise training is known as an effective intervention method in the treatment of rotator cuff/subacromial impingement problems, there is no definite consensus on which type of exercise is more effective. However, when previous literature studies from 2022 were examined, a single pilot study was found that examined the effect of specific slow resistance training on symptoms in rotator cuff tendinopathy; No studies could be found comparing specific slow slow resistance training with other exercise interventions. The aim of this thesis, which the investigators planned in the light of this information, is to analyze and compare the effects of heavy slow resistance training and eccentric exercise training on pain, function, supraspinatus tendon structure, muscle strength, range of motion, subjective perception of improvement and treatment satisfaction in individuals with subacromial shoulder pain associated with rotator cuff tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Describing subacromial pain
* Rotator cuff tendinopathy (subacromial impingement syndrome, biceps tendinitis and rotator cuff I. and II. stage diagnosis)
* Continuation of diagnostic symptoms for at least 30 days

Exclusion Criteria:

* Prior shoulder surgery
* Sign of cervical radiculopathy
* Shoulder instability or history of upper extremity fracture
* Full-thickness rotator cuff tear
* Adhesive capsulitis
* Humeroscapular periarthritis (osteoarthritis, inflammatory arthropathies, etc.)
* Neoplasm/malignant status
* Other independent from shoulder problem being on regular analgesic therapy for ongoing painful conditions
* Subacromial corticosteroids in the last 2 months having received an injection or participating in a shoulder rehabilitation program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The supraspinatus tendon thickness and elasticity | 6 weeks
  Affected party the supraspinatus tendon thickness and elasticity value will be evaluated by shear-wave elastography by a specialist radiologist.

SECONDARY OUTCOMES:
Isometric muscle strength | 6 weeks
  Isometric muscle strength of the external and internal rotators of the shoulder and the supraspinatus muscle will be evaluated by manual muscle testing. For manual muscle testing a digital hand-held dynamometer will be used.
Shoulder range of motion | 6 weeks
  A digital inclinometer will be used to evaluate the range of motion of the shoulder joint. Reviews shoulder flexion, abduction, internal and external rotation movements will be done. Active movement without pain (painless NEH) will be measured. All measurements will be repeated three times and averaged and recorded in degrees.
The level of pain and disability associated with the shoulder | 6 weeks
  The Shoulder Pain And Disability Index (SPADI), to assess the level of shoulder-related pain and disability will be used.
Shoulder pain severity | 6 weeks
  The Numerical Pain Rating Scale will be used to assess the severity of shoulder pain.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Ha Esen, PhD. c, Principal Investigator — Gazi University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- Gazi University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beyer R, Kongsgaard M, Hougs Kjaer B, Ohlenschlaeger T, Kjaer M, Magnusson SP. Heavy Slow Resistance Versus Eccentric Training as Treatment for Achilles Tendinopathy: A Randomized Controlled Trial. Am J Sports Med. 2015 Jul;43(7):1704-11. doi: 10.1177/0363546515584760. Epub 2015 May 27. PMID 26018970
- [Background] Bateman M, Adams N. A randomised controlled feasibility study investigating the use of eccentric and concentric strengthening exercises in the treatment of rotator cuff tendinopathy. SAGE Open Med. 2014 Jan 28;2:2050312113520151. doi: 10.1177/2050312113520151. eCollection 2014. PMID 26770702
- [Background] Macias-Hernandez SI, Garcia-Morales JR, Hernandez-Diaz C, Tapia-Ferrusco I, Velez-Gutierrez OB, Nava-Bringas TI. Tolerance and effectiveness of eccentric vs. concentric muscle strengthening in rotator cuff partial tears and moderate to severe shoulder pain. A randomized pilot study. J Clin Orthop Trauma. 2020 Aug 3;14:106-112. doi: 10.1016/j.jcot.2020.07.031. eCollection 2021 Mar. PMID 33680816
- [Background] Schydlowsky P, Szkudlarek M, Madsen OR. Comprehensive supervised heavy training program versus home training regimen in patients with subacromial impingement syndrome: a randomized trial. BMC Musculoskelet Disord. 2022 Jan 15;23(1):52. doi: 10.1186/s12891-021-04969-0. PMID 35033043